CLINICAL TRIAL: NCT04972240
Title: Evaluation of Stability, Marginal Bone Loss and Occlusal Load Analysis of Customized Posterior Hybrid PEEK Abutments Supported by Short Implants
Brief Title: Stability, Marginal Bone Loss and Occlusal Load Analysis of PEEK Abutment Supported on Short Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Shahenda Tarek Abu Amu, assistant lecture, Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P-CR-21-03
Record Dates: First submitted 2021-07-15; First posted 2021-07-22 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Marginal Bone Loss and Loss of Osteointegration of Short Implant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Customized PEEK abutment/ crown on a Ti base. (Active Comparator)
  Interventions: Other: customization of abutment
- Prefabricated titanium abutment, supporting ceramometal separate crown. (No Intervention)

INTERVENTIONS:
Other: customization of abutment — we will customize abutment for every patient not ready made
  Arms: Customized PEEK abutment/ crown on a Ti base.

SUMMARY:
this study will be directed toward evaluating stability, marginal bone loss and occlusal load of posterior customized PEEK abutments on Ti-bases supported by short implant

DETAILED DESCRIPTION:
although short implant solved many clinical problems; it is sometimes associated with loss of osseointegration which is firstly expressed by peri-implantitis and marginal bone loss. Also, PEEK is a very promising material characterized by low modulus of elasticity thus it can act as a shock absorber. Whether constructing superstructure components of short implant from PEEK will improve their performance or not is lacking in the dental literature.

To conduct the present study, the following will be used:

1. Customized screw retained PEEK abutment/crown on a Ti base.
2. Prefabricated titanium abutment.
3. Short implant. The study will be conducted on 12 patients with missing single posterior tooth indicated for short implants) near anatomical structure or atrophic ridge), attending the outpatient clinic of the Crowns and Bridges department, Faculty of Dental Medicine for Girls, Al-Azhar University.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range of patients 30-45 years old, with no gender prediction, able to read and sign the informed consent. 2. Patient with missing posterior tooth indicated for replacement with short implant as there are any anatomical limitation (near maxillary sinus or inferior alveolar nerve) or atrophic ridge. 3. Opposing natural teeth should be present. 4. The edentulous ridge should be free from any infection or remining root. 5. Patient should be able to tolerate surgical procedure of implant procedures physically and psychologically. 6. Patient should be willing to return for follow-up examination and evaluation.

Exclusion Criteria:

* 1. Patients with active periodontal diseases. 2. Patient with poor oral hygiene and motivation. 3. Pregnant women. 4. Patient with unrealistic expectations. 5. Patients with parafunctional habits and smoker. 6. Patient with systemic disease and immunocompromised patients which will prevent surgical procedure. 7. Recent extraction or extraction socket with infection or remining root.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
decrease marginal bone loss around short implant | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Alazhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes